CLINICAL TRIAL: NCT02359630
Title: The EasyTube® in General Anesthesia: A Multicenter Study Comparing EasyTube and Endotracheal Tube
Brief Title: Multicenter Study of EasyTube® Compared to Endotracheal Tube in General Anesthesia
Acronym: EasyTube
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Frass, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2015-01-18; First posted 2015-02-10 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Airway Morbidity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EasyTube (Active Comparator): Use of EasyTube during general anesthesia
  Interventions: Device: EasyTube; Device: Endotracheal tube
- Endotracheal tube (Experimental): Use of endotrachel tube during general anesthesia
  Interventions: Device: EasyTube; Device: Endotracheal tube

INTERVENTIONS:
Device: EasyTube — Insertion for ventilation
Device: Endotracheal tube — Insertion for ventilation

SUMMARY:
Evaluation of the EzT in comparison with the endotracheal tube (ETT) for its use during general anesthesia.

DETAILED DESCRIPTION:
There is a recent paper suggesting that general anesthesia with the EzT is feasible and by no means worse than anesthesia with a conventional ETT, and there is little but growing evidence that narcosis with this SAD can be continued during general anesthesia. This brings up several potential benefits: The larger balloons of the EzT are less traumatic to the mucosal tissue compared to a conventional ETT or to a laryngeal mask. Since the insertion of the EzT can be performed without using a laryngoscope, this also reduces tissue damage and tooth injuries caused by a laryngoscope. Also, It has been demonstrated that a similar SAD - the Combitube - can be placed by anesthesiologists with relatively little formal training and that ventilation during elective surgery is feasible. However, such detailed data are missing for the EzT, with only smaller, monocenter-studies available. The next logical step was therefore to systematically evaluate the EzT beyond its purpose as a rescue device in a prospective, randomized multicenter-study to evaluate the use of the EzT in comparison with the ETT during general anesthesia.

Methods 400 patients with ASA status I-II scheduled for elective surgery in 4 centers were randomized to either the EzT group (n=200) or the ETT group (n=200).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II and were scheduled for an elective surgery requiring general anesthesia

Exclusion Criteria:

* Age < 18 years
* Acute or chronic lung disease
* Patients presenting with sore throat
* Known esophageal disease
* Oropharyngeal abnormalities
* Patients with a cervical spine disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
success of insertion | 60 seconds
  success of insertion

SECONDARY OUTCOMES:
duration of ventilation | 60 seconds
  Recording of duration of ventilation, inspiratory and expiratory minute volumes, oropharyngeal leak pressure, and rate of complications
inspiratory and expiratory minute volumes | 60 seconds
  minute volumes recorded during inspiration or expiration
oropharyngeal leak pressure | 60 seconds
  pressure exerted by the inflatable cuff/balloon on the pharyngeal wall
rate of complications | 60 seconds
  injury to the mucosa of the mouth, nose, etc.
rating of insertion difficulty | 60 seconds
  Anesthesiologists describe the difficulty of insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Result] Gaitini LA, Vaida SJ, Mostafa S, Yanovski B, Croitoru M, Capdevila MD, Sabo E, Ben-David B, Benumof J. The Combitube in elective surgery: a report of 200 cases. Anesthesiology. 2001 Jan;94(1):79-82. doi: 10.1097/00000542-200101000-00016. PMID 11135725